CLINICAL TRIAL: NCT02926612
Title: Pathogen Identification in Pediatric Hematopoietic Stem Cell Transplant Patients With Suspected Lower Respiratory Tract Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pediatric Blood and Marrow Transplant Foundation, Inc. (Other)
Collaborators: St. Baldrick's Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SUP1601
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Lower Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HCT recipients ages ≤21 years: HCT recipients ages ≤21 years for whom lower respiratory secretions are being collected for direct patient care.
  Interventions: Other: Next Generation Genomic Sequencing

INTERVENTIONS:
Other: Next Generation Genomic Sequencing — DNA and RNA are extracted from biospecimens, amplified, sequenced, and then compared to known microbe databases, allowing for quantitative identification of non-host organisms

SUMMARY:
This is a multicenter prospective collection of leftover respiratory tract secretions, paired blood and NP swabs, and clinical circumstances from pediatric HCT patients, followed by next generation genomic sequencing, transcriptome analysis, protein biomarker measurement, and statistical modeling.

DETAILED DESCRIPTION:
This study is a multicenter cross-sectional observational analysis of unused lower respiratory tract secretions collected from children with a history of HCT who are undergoing evaluation for pulmonary complications. Patients will be screened and enrolled by study coordinators at each site, who will collect and submit biospecimens as well as patient characteristics and clinical outcomes. Metagenomic NGS will be performed on these biospecimens in an attempt to identify microbial pathogens and markers of host response to infection, including immune activation, inflammation, and cell damage. This study will then correlate these results with patient characteristics, clinical microbiology test results, and clinical outcomes in order to evaluate the utility of metagenomics NGS in improving the diagnosis of LRTI in our pediatric HCT population.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be ≤21 years of age with a history of HCT of any type at any point in the past, and are planned to undergo clinically-indicated collection of any lower respiratory specimen, including but not limited to bronchoalveolar lavage (either via a plugged telescoping catheter such as a CombiCath, or with fiberoptic bronchoscopy) and tracheal aspirate.
* For the purposes of this study, induced or spontaneous sputum is not considered a lower respiratory tract specimen.
* Patients may have any underlying indication for clinical testing of lower respiratory secretions, including but not limited to suspected infection, non-infectious inflammation, obstructive or restrictive lung disease, pulmonary edema, pleural effusions, alveolar hemorrhage, aspiration, or pulmonary vascular disease.
* Patients who have not undergone HCT but plan to undergo HCT in the future, hereafter referred to as pre-HCT patients, may also be enrolled.
* Pre-HCT patients must have intention to undergo stem cell transplantation in the future and include but are not limited to patients with primary immunodeficiency, patients with malignancy undergoing induction or consolidation chemotherapy, and HCT patients with selected cell sources who are undergoing pre-transplant conditioning but have not yet received their cellular infusion.

Exclusion Criteria:

* Patients will not be >21 years of age.
* Patients who do not have a clinical indication for obtaining lower respiratory secretions for testing as part of their direct patient care will be excluded.
* Patients who do not have sufficient respiratory secretions remaining after collection and aliquoting for indicated clinical tests ordered by the treating clinician will also be excluded.
* Patients who undergo lower respiratory testing solely to evaluate for relapsed malignancy will be excluded.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HCT recipients ages ≤21 years for whom lower respiratory secretions are being collected for direct patient care.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate and quantify the utility of NGS in improving the diagnosis of LRTI in pediatric HCT patients. | 3 years

SECONDARY OUTCOMES:
Evaluate the utility of human gene expression profiling in improving our understanding of host-microbe interactions in infectious and alloreactive pulmonary inflammation. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Zinter, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient results will be available to the patient site, but it is undecided whether or not to make these results available to everyone.